CLINICAL TRIAL: NCT00497263
Title: End-to-End Compression Anastomosis for Left-sided Colectomy Endo-CAR Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Niti Medical Technologies Ltd. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: CLP-43-01 Rev 01
Record Dates: First submitted 2007-07-04; First posted 2007-07-06 (Estimated); Last update posted 2011-06-29 (Estimated); Status verified 2011-06

CONDITIONS: Colorectal Cancer; Diverticulitis
MeSH Terms: conditions — Colorectal Neoplasms; Diverticulitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Niti CAR

SUMMARY:
the purpose of this study is to evaluate the safety and effectiveness of the Niti CAR-device in the creation of colorectal anastomosis

ELIGIBILITY:
Inclusion Criteria:

* Patient age over 18
* Patient schedule for colonic surgery requiring E-t-E anastomosis
* Patient is able to understand and to sign the Informed Consent Form

Exclusion Criteria:

* Patient has known allergy to Nickel
* Patient with bowel obstruction, strangulation, peritonitis, perforation, local or systemic infection
* Patient on regular steroid medication
* Patient with preexisting sphincter problems or evidence of extensive local disease of the pelvis
* Patient following radiation (that compromised the anastomosis)
* Patient who are undergoing a defunctioning stoma
* Patient with contraindication to general anesthesia
* Patient who is currently participating in other clinical trial
* Patient who refuse consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
functioning anastomosis & no occurrence of adverse events related to device use | during hospitalization and until 3 months after discharge

CONTACTS AND LOCATIONS:
Overall Officials: André D'Hoore, MD, PhD, Principal Investigator — University Hospitals Gasthuisberg Leuven
Locations (1):
- University Hospitals Gasthuisberg Leuven, Leuven, Brabant, Belgium